CLINICAL TRIAL: NCT06661356
Title: Determining the Impact of Peer-led Community-based PrEP Delivery Among Youth in Brazil: A Randomized Controlled Trial
Brief Title: Peer-led Community-based PrEP Delivery Among Youth in Brazil
Acronym: COMPrEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Sao Paulo (Other); Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Katia J. Bruxvoort, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-300013551; 1R01MH135769-01A1 (NIH)
Record Dates: First submitted 2024-10-18; First posted 2024-10-28 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Pre-Exposure Prophylaxis (PrEP); HIV
Keywords: PrEP; Pre-Exposure Prophylaxis; HIV; Peer lay workers; Youth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding will not be possible for participants, peer lay workers, and health providers, but the data management and analysis teams will be blinded to the study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Arm (No Intervention): Participants randomized to the standard care arm will receive PrEP at a health facility from a physician or nurse.
- COMPrEP Intervention (Experimental): Participants randomized to the COMPrEP intervention will receive PrEP from peer lay workers at private community locations.
  Interventions: Behavioral: COMPrEP

INTERVENTIONS:
Behavioral: COMPrEP — Participants will be paired with peer lay workers and will meet with peer lay workers at private community location. They will discuss options for oral PrEP with peer lay workers and be provided provide daily oral PrEP or event-driven (2-1-1) PrEP. Participants will take part in rapid HIV testing at each visit. They will also meet with peer lay workers at private community location for follow-up at 1, 5, 9, and 13 months.
  Arms: COMPrEP Intervention

SUMMARY:
The goal of this project is to conduct a series of studies to refine, test, and understand experiences with a peer-led community-based intervention in which youth will be integrated into health care teams and trained to deliver HIV pre-exposure prophylaxis (PrEP) to their peers. The study team will conduct a randomized trial to determine if peer delivery of PrEP to youth aged 15-24 in Brazil will increase PrEP uptake, persistence, and adherence compared to standard PrEP care provided in health facilities.

DETAILED DESCRIPTION:
HIV is declining in many parts of the world, but rising in Latin America, including Brazil. The HIV epidemic in Brazil, including the number of new infections, is concentrated among youth aged 15-24. Youth in Brazil face obstacles to HIV prevention. Use of HIV pre-exposure prophylaxis (PrEP) lags far behind PrEP need in Brazil. There is international momentum to promote PrEP as prevention and to increase access to low barrier care. Peer lay workers are a promising approach to address the unmet need for PrEP uptake and adherence among youth in Brazil.

COMPrEP is a multi-site randomized controlled trial designed to determine if peer delivery of PrEP to youth aged 15-24 in Brazil will increase PrEP uptake, persistence, and adherence compared to standard PrEP care provided in affirming health facilities. Eligible youth (N=1400) in two municipalities in Brazil (i.e., Salvador and São Paulo) will be randomized to 1:1 to either the COMPrEP intervention arm (PrEP access through peer lay workers in community venues) or the standard care arm (PrEP access through health providers at health facilities). It is anticipated that approximately 245 and 140 youth will initiate PrEP in intervention and standard care arms, respectively, and these will be followed for 12 months, facilitating measurement of PrEP adherence and persistence outcomes on this subset.

ELIGIBILITY:
Eligibility Criteria:

* Aged 15-24 years
* Candidate for HIV prevention
* Sexually active
* Not currently using PrEP
* Willing to discuss oral PrEP
* Agree to be randomized to either intervention or standard care arm

Exclusion Criteria:

* HIV positive test result
* Not currently sexually active
* Currently using PrEP

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1400 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
PrEP Uptake | Within 1 month of enrollment
  Received at least one PrEP prescription

SECONDARY OUTCOMES:
PrEP Adherence Biomarker | 1 month
  Positive point of care urine tenofovir assay
PrEP Adherence Self-Report | At 1, 5, 9, and 13 months
  Number of pills taken in the past 30 days
PrEP Persistence | 5 months and 13 months
  Continuing to take PrEP at 5 months and 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Katia J Bruxvoort, PhD, Principal Investigator — University of Alabama at Birmingham School of Public Health
Locations (2):
- Brazil (2):
  - Federal University of Bahia, Salvador, Estado de Bahia
  - University of São Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with anyone outside of the study team.